CLINICAL TRIAL: NCT04902417
Title: Influence of Increased Dairy Product Consumption on Markers of Inflammation and Cardiometabolic Disease
Brief Title: Dairy and Inflammation Study
Acronym: DRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Andrea Josse, Assistant Professor, York University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-177
Record Dates: First submitted 2021-05-11; First posted 2021-05-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inflammation; Overweight and Obesity; Cardiometabolic Risk
Keywords: Dairy; Diet; Inflammation; postprandial
MeSH Terms: conditions — Inflammation; Overweight; Obesity | interventions — Yogurt; Cheese; Milk

STUDY DESIGN:
Intervention Model Description: Two-phase, randomized, controlled, crossover trial design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dairy Habitual Diet (No Intervention): Participants will follow their usual diet for 6-weeks, which includes low dairy consumption as screened for with the inclusion criteria.
- High Dairy Diet (Experimental): Participants will be provided with 3 servings of dairy per day to replace other foods within their diet (preventing weight gain over the intervention period) for 6-weeks
  Interventions: Other: Dairy Foods (Yoghurt, Cheese, Milk)

INTERVENTIONS:
Other: Dairy Foods (Yoghurt, Cheese, Milk) — Participants will be provided with a combination of dairy products (Yoghurt, Cheese, Milk) to be consumed daily, for a total of 3 servings per day
  Arms: High Dairy Diet

SUMMARY:
The purpose of this study is to determine whether 6-weeks of increased dairy consumption can reduce inflammation and other markers of chronic disease while fasted or following a high-fat meal.

DETAILED DESCRIPTION:
Following the acquisition of informed consent, eligibility to participate in the study will be determined using questionnaires, and certain parameters determined from a finger-prick blood sample. Eligible participants will be assigned to complete two 6-week dietary interventions in random order, with at least a 4 week "wash out" period (i.e. their habitual eating) in between. The two dietary interventions are: 1) Participants normal, low-dairy diet; and 2) A higher dairy diet where 3 servings per day of dairy foods are provided. Prior to beginning either 6-week diet intervention, participants will be asked to attend the laboratory at York University after an overnight fast to undergo baseline testing.

Following baseline testing, participants will meet with a registered dietitian (RD) to discuss each diet arm. Specifically, if they are on the dairy diet, participants will receive advice on how to incorporate these dairy foods into their diet by replacing other foods of similar energy content so as to not increase their total energy intake and body weight. They will meet with the RD at several other times throughout the study. During each 6-week diet period, they will be asked to keep their physical activity levels constant and to not adopt any other major dietary changes during the study.

At the end of each 6-week intervention period, participants will be asked to return to York University to repeat the initial set of tests performed at baseline. In addition to the fasted tests, a number of tests will be performed after asking participants to consume a high-fat test meal (i.e. a fast-food breakfast). Various measurements will continue to be taken for around 6 hours after this meal is consumed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 25 kg/m2
* ≤ 2 structured exercise sessions/week
* Habitual low dairy consumption (≤ 1 serving/day)
* Having at least two other metabolic risk factors based on clinical guidelines:

  * Elevated blood pressure (≥130/≥85 mm Hg)
  * Impaired fasting glucose (≥5.6 mmol/L) measured using a finger prick sample
  * Impaired fasting triglycerides (≥1.7 mmol/L) or high-density lipoprotein (<1.03 mmol/L for males, <1.3 mmol/L for females) measured using a finger prick blood sample.
  * Increased waist circumference (≥102 cm for males and ≥88 cm for females).
  * Borderline high fasting low-density lipoprotein (≥3.5 mmol/L) or total cholesterol (≥5.2 mmol/L).

Exclusion Criteria:

* Allergy to dairy foods, diagnosed lactose intolerance or an aversion to foods provided during the study
* Previous history of diabetes and/or related cardiovascular disease
* The use of multiple medications for managing lipids, glucose and/or blood pressure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Fasting Inflammation | pre-intervention
  Concentration of Interleukin-6
Fasting Inflammation | immediately after the 6 week intervention
  Concentration of Interleukin-6
Postprandial Inflammation | 1 hour post meal
  Concentration of Interleukin-6
Postprandial Inflammation | 2 hour post meal
  Concentration of Interleukin-6
Postprandial Inflammation | 3 hour post meal
  Concentration of Interleukin-6
Postprandial Inflammation | 4 hour post meal
  Concentration of Interleukin-6
Postprandial Inflammation | 5 hour post meal
  Concentration of Interleukin-6

SECONDARY OUTCOMES:
Fasting Lipids | pre-intervention
  Concentration of serum cholesterol
Fasting Lipids | immediately after the 6 week intervention
  Concentration of serum cholesterol
Fasting Lipids | pre-intervention
  Concentration of serum triglycerides
Fasting Lipids | immediately after the 6 week intervention
  Concentration of serum triglycerides
Fasting glucose | pre-intervention
  Concentration of blood glucose
Fasting glucose | immediately after the 6 week intervention
  Concentration of blood glucose
Fasting insulin | pre-intervention
  Concentration of blood insulin
Fasting insulin | immediately after the 6 week intervention
  Concentration of blood insulin
vascular measures | pre-intervention
  flow-mediated dilation (FMD)
vascular measures | immediately after the 6 week intervention
  flow-mediated dilation (FMD)
Body composition | pre-intervention
  fat mass (kg)
Body composition | immediately after the 6 week intervention
  fat mass (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Skelly, PhD, Study Director — York University; Joel Prowting, MSc, Study Director — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prowting JL, Fraschetti EC, Pereira TJ, Tucker JA, Gagnon S, Cheng N, Edgell H, Wright DC, Klentrou P, Perry CG, Josse AR. Inflammatory Cytokine Responses to 6 Wks of Increased Dairy Intake in Individuals with Overweight and Obesity-A Randomized Crossover Trial. J Nutr. 2026 Jan;156(1):101227. doi: 10.1016/j.tjnut.2025.10.040. Epub 2025 Oct 30. PMID 41176279